CLINICAL TRIAL: NCT03209349
Title: Investigation of Cecal Intubation Rates and Pain Levels Between Water Exchange and Air Insufflation Flexible Sigmoidoscopy: A Randomized Controlled Study
Brief Title: Investigation of Cecal Intubation Rates and Pain Levels Between Water Exchange and Air Insufflation Flexible Sigmoidoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kelowna Gastroenterology Associates (Other)
Collaborators: Veteran Affairs Sepulveda Ambulatory Care Cente (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 2016-17-078-I
Record Dates: First submitted 2017-06-14; First posted 2017-07-06 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer
Keywords: Sigmoidoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study interviewer and the patient will be blinded to the procedure type both during and following the procedure type both during and following the procedure by concealing the monitors and relevant equipment from their sight.
  The physician performing the procedure will be blinded to the procedure type until the patient is brought into the procedure room. They will open the allocation envelope once the patient has been placed and positioned on the procedure bed.
  Neither the patient, the RN, nor the research assistant, who will be conducting the follow-up interviews, will be informed of the study arm. Patient assignment will be managed by the study project manager and will be kept in a password protected file and will remain separate from other study data until the time of the final analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water Exchange Sigmoidoscopy (Experimental): As per standard practices, the patient will be walked to the procedure room and positioned in the left lateral position on the procedure bed, without pre-operative anesthesia. The procedures will be completed within the ambulatory endoscopy clinic at Kelowna General Hospital. The study will use the same colonoscopes that are already being used at KGH for colonoscopy. These are the Olympus 190 series colonoscopes. They can and will be fitted to support both water and air exchange.
  For patients assigned the water exchange intervention arm, the insertion of the scope will be followed by infusion and suction of water to minimally distend the lumen. If the lumen does not open, the instrument will be retracted slightly and the infusion started again. As the scope is inserted and progressed through the intestinal lumen some of the infused water will be suctioned back constantly, exchanging clean for opaque water.
  Interventions: Procedure: Water Exchange Sigmoidoscopy
- Air Insufflation Sigmoidoscopy (Active Comparator): As per standard practices, the patient will be walked to the procedure room and positioned in the left lateral position on the procedure bed, without pre-operative anesthesia. The procedures will be completed within the ambulatory endoscopy clinic at Kelowna General Hospital. The study will use the same colonoscopes that are already being used at KGH for colonoscopy. These are the Olympus 190 series colonoscopes. They can and will be fitted to support both water and air exchange.
  For patients assigned to the air insufflation intervention arm, extended sigmoidoscopy will be performed with the minimum insufflation required to reach the cecum.
  Interventions: Procedure: Air Insufflation Sigmoidoscopy

INTERVENTIONS:
Procedure: Water Exchange Sigmoidoscopy — See arm description.
  Arms: Water Exchange Sigmoidoscopy
Procedure: Air Insufflation Sigmoidoscopy — See arm description.
  Arms: Air Insufflation Sigmoidoscopy

SUMMARY:
This study evaluates how often patients without sedation that receive screening sigmoidoscopy are able to have their full colon examined without significant discomfort by comparing a new colonoscopy technique known as the water exchange technique to the traditional air insufflation technique. It compares the differences between complete colon exam rates for water exchange when compared to the traditional air technique. Patients will be randomised and blinded to the procedure type.

Previous studies have shown that the water exchange method is associated with a significant reduction in discomfort and often allows patients to receive colonoscopy without sedation or with only minimal sedation. However, the potential for water exchange to be used in the screening setting has yet to be evaluated. As per standard practices in sigmoidoscopy screening, patients will not be sedated. However, unlike standard practices in sigmoidoscopy screening, while maintaining minimal levels of discomfort, the investigators will attempt to scope beyond the distal colon.

DETAILED DESCRIPTION:
Purpose:

This study is being conducted to evaluate whether a new technique, known as the water exchange technique can more frequently allow for the full colon to be examined in patients undergoing screening sigmoidoscopy.*

Hypothesis & Goals & Objectives:

It is hypothesised that there will be a 20% or greater difference in cecal intubation rate (ability for the colonoscope to reach the Ileocecal juncture, and thereby provide full examination of the colon) at a minimal and acceptable level of discomfort in non-sedated colon screening patients receiving a scope using the water-exchange method, when compared to the air insufflation method.

Justification:

Previous studies have shown that the water exchange method is associated with a significant reduction in discomfort and often allows patients to receive colonoscopy without sedation or with only minimal sedation. The ability to increase the likelihood of full colon examination at minimal discomfort has the opportunity to improve upon screening practices and increase the likelihood of patient participation as discomfort and fear of discomfort is a major factor that limits uptake of sigmoidoscopy and colonoscopy screening.

Research Design:

This study takes a patient and interviewer blinded and randomised study design. Patients will be randomly assigned to receive either the water exchange method or the air insufflation method. Rates of cecal intubation are compared across study arms.

Statistical Analysis Plan:

Effect differences in cecal intubation rates, and responses to whether the scope that they received was more uncomfortable than they expected, and whether they would be willing to receive the test again at their next screening interval will be compared using the Chi-Squared or, when the data necessitates, Fisher's Exact Test. Assuming a non-normal distribution in reported pain scores, the Mann Whitney U test will be used to assess the differences in maximum reported pain according to the Wong Baker Faces Pain Rating Scale between study arms.

*The term sigmoidoscopy is used here as patients are prepared for the procedure using a standard sigmoidoscopy protocol, rather than colonoscopy. That is, sedation is not administered; this is a standard practice for sigmoidoscopy procedures but not for colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic average risk (as per BC colon screening guidelines) individuals
* Ages 50-74 years of age

Exclusion Criteria:

* A sigmoidoscopy or colonoscopy within 10 years,
* A FIT within 2 years,
* Individuals classified with any high-risk screening criteria in accordance to the

BC colon screening guidelines including:

* a personal history of adenoma,
* a first degree relative that was diagnosed with colorectal cancer or multiple adenomas under the age of 60,
* two or more first degree relatives with colorectal cancer at any age, longstanding inflammatory bowel diseases,
* a family history of familial adenomatous polyposis or hereditary nonpolyposis colorectal cancer, - Individuals presenting with rectal pain, rectal bleeding, abdominal pain, or unintentional weight loss at the time of the examination.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Full colon exam | Immediately following the procedure
  Ability for patient to receive full exam of the colon with minimal discomfort

SECONDARY OUTCOMES:
Recalled Discomfort | Immediately following the procedure
  Patient will be contacted at 24 hours following the procedure and in order to document whether the scope was more uncomfortable than expected and if the patient would be willing to receive the test again at their next screening interval.
Adenoma detection rates | Immediately following the procedure
  Histopathological testing and reporting will follow standard practices and adenoma detection rates will be documented and compared between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Perini, MD, Principal Investigator — Kelowna General Hospital, Department of Gastroenterology; Adrian Bak, MD, Principal Investigator — Kelowna General Hospital, Department of Gastroenterology
Locations (2):
- Sepulveda Ambulatory Care Center, North Hills, California, United States
- Brent Parker, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No